CLINICAL TRIAL: NCT02248090
Title: Phase I, Open-Label, Multicentre Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumour Activity of Ascending Doses of AZD9496 in Women With Estrogen Receptor Positive HER-2 Negative Advanced Breast Cancer
Brief Title: AZD9496 First Time in Patients Ascending Dose Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D6090C00001
Record Dates: First submitted 2014-09-22; First posted 2014-09-25 (Estimated); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: ER+ HER2- Advanced Breast Cancer
Keywords: Phase 1; Safety; Tolerability; Pharmacokinetics; Ascending Doses; Estrogen Receptor Positive; Her2 Negative; Advanced Breast Cancer
MeSH Terms: interventions — AZD9496

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD9496 (Experimental): AZD9496 dose escalation and expansion(s)
  Interventions: Drug: AZD9496

INTERVENTIONS:
Drug: AZD9496 — AZD9496
Drug: AZD9496 — If initial dosing of AZD9496 is tolerated then subsequent cohorts will test increasing doses until a maximum tolerated dose or maximum feasible dose is defined

SUMMARY:
This is a phase 1 open label multicentre study of AZD9496 administered orally in patients with advanced ER+ HER2 negative breast cancer. The study design allows an escalation of dose with intensive safety monitoring to ensure the safety of patients. The study will determine the maximum tolerated dose. In addition, expansion cohort(s) at potential therapeutic dose(s) in patients with or without ESR1 mutations will be enrolled to further determine the safety, tolerability, pharmacokinetics and biological activity of AZD9496

DETAILED DESCRIPTION:
A Phase I, Open-Label, Multicentre Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumour Activity of Ascending Doses of AZD9496 in Women with Estrogen Receptor Positive HER-2 Negative Advanced Breast Cancer

ELIGIBILITY:
Inclusion Criteria: Provision of signed and dated, written informed consent prior to any mandatory study specific procedures, sampling and analyses. Aged at least 18 years. Any menopausal status. Pre- or peri-menopausal women must have commenced treatment with an LHRH agonist at least 4 weeks prior to starting study treatment and must be willing to continue to receive LHRH agonist therapy for the duration of the trial. Histological or cytological confirmation of adenocarcinoma of the breast. ER-positive according to local laboratory; HER-2 negative. Metastatic disease or locoregionally recurrent disease which is not amenable to treatment with curative intent. Disease progression after at least 6 months of endocrine therapy for ER+ breast cancer. Radiological or objective evidence of progression on or after the last systemic therapy prior to starting study treatment. Receipt of ≤2 lines of prior chemotherapy for advanced disease. Females of child-bearing potential must agree to use adequate contraceptive measures, must not be breast feeding and must have a negative pregnancy test prior to start of dosing. Eastern Cooperative Oncology Group (ECOG) performance status 0-1 with no deterioration over the previous 2 weeks and minimum life expectancy of 12 weeks.

Exclusion Criteria: Any cytotoxic chemotherapy, investigational agents or other anti-cancer drugs for the treatment of advanced breast cancer from a previous treatment regimen or clinical study within 14 days of the first dose of study treatment. Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 at the time of starting study treatment with the exception of alopecia. Presence of life-threatening metastatic visceral disease, uncontrolled central nervous system metastatic disease or symptomatic pulmonary lymphangitic spread. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension, active bleeding diatheses, or active infection. Unexplained symptomatic endometrial disorders. Uncontrolled symptomatic thyroid dysfunction. Inadequate bone marrow reserve or organ function

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-10-22 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2019-04-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | Routine safety assessments, throughout the period that patients receive AZD9496 up to 28 days following discontinuation of last dose of study treatment.
  Safety and tolerability in terms of adverse events, serious adverse events (including death) and safety measures: ECG, physical examination, vital signs and laboratory variables. Definition of maximum tolerated dose (MTD) or maximum feasible dose (MFD) by measuring the number of evaluable patients with dose-limiting toxicities.Time frame DLT period 28 days

SECONDARY OUTCOMES:
Single and multiple dose pharmacokinetics of AZD9496 | 12 weeks
  measurement of plasma levels of AZD9496 at pre-defined intervals in order to establish pharmacokinetic parameters
4β-hydroxycholesterol concentration in blood | 12 weeks
  Understanding of the CYP3A4 induction potential of AZD9496 by measuring 4β-hydroxycholesterol concentration in blood samples at pre-defined intervals
Antitumour activity | every 8 weeks for 24 weeks and then every 12 weeks thereafter until disease progression
  Antitumour activity by evaluation of tumour response assessments using Response Evaluation Criteria in Solid Tumours (RECIST 1.1)

CONTACTS AND LOCATIONS:
Overall Officials: Erika Hamilton, Principal Investigator — Nashville Hospital, United States; Justin Lindemann, Study Director — AstraZeneca
Locations (6):
- United States (3):
  - Florida Cancer Specialists, Sarasota, Florida
  - Research Site, New York, New York
  - Sarah Cannon, Nashville, Tennessee
- Seoul National Univ. Hospital, Seoul, South Korea
- United Kingdom (2):
  - Research Site, Cambridge
  - Christie, Manchester